## PROTOCOL TITLE

Cerebellar transcranial magnetic stimulation (TMS) in psychotic disorders: effect on time perception, executive function, and mood and psychotic symptoms

NCT Number: NCT02642029

**Date:** August 22, 2022

## Statistical Analyses:

We will test for group differences in demographic and clinical variables using  $\chi^2$  and t-tests or ANOVA, as appropriate. To examine the effect of TBS conditions on symptoms (as measured by visual analog scale scores, which are not normally distributed), we will conduct the non-parametric Friedman's test. For all other outcome measures, we will use mixed model regressions with TMS condition (cTBS, iTBS, or sham TBS), time (pre-TMS, post-TMS), and the interaction of condition x time as the primary variables of interest. To test the association between performance on the interval discrimination task (IDT) and symptoms, we will run mixed model regression models with TMS condition and time in addition to symptom score as the primary variable of interest.